CLINICAL TRIAL: NCT04128293
Title: A Randomized, Open-Label, Single Dose, Four-Period Crossover Clinical Trial to Assess the Relative Bioavailability of a Tablet Compared to a Capsule of GSK3640254 and to Assess the Effect of Food on the GSK3640254 Tablet in Healthy Participants
Brief Title: A Relative Bioavailability and Food-Effect Study of GSK3640254 Tablet and Capsule Formulations in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: GSK investigating manufacturing site malfunction and assessing impact; Study 209713 Early Terminated due to risk of potential contamination of study tablets.
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 209713
Record Dates: First submitted 2019-10-01; First posted 2019-10-16 (Actual); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: Healthy participants; GSK3640254; Human immunodeficiency virus (HIV); Safety
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — GSK3640254

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to 1 of 4 treatment sequences (ABCD, BADC, CDAB, or DCBA) in each treatment period.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 - Treatment ABCD (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment A- Reference), capsules, orally under moderate fat conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment B- Test), tablets, orally under moderate fat conditions on Day 1 in second intervention period; followed by GSK3640254 200 mg (Treatment C- Reference), tablets, orally under fasted conditions on Day 1 in third intervention period; further followed by GSK3640254 200 mg (Treatment D- Test), tablets, orally under high fat conditions on Day 1 in fourth intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet; Drug: GSK3640254 Capsule
- Sequence 2 - Treatment BADC (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment B- Test), tablets, orally under moderate fat conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment A- Reference), capsules, orally under moderate fat conditions on Day 1 in second intervention period; followed by GSK3640254 200 mg (Treatment D- Test), tablets, orally under high fat conditions on Day 1 in third intervention period; further followed by GSK3640254 200 mg (Treatment C- Reference), tablets, orally under fasted conditions on Day 1 in fourth intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet; Drug: GSK3640254 Capsule
- Sequence 3 - Treatment CDAB (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment C- Reference), tablets, orally under fasted conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment D- Test), tablets, orally under high fat conditions on Day 1 in second intervention period; followed by GSK3640254 200 mg (Treatment A- Reference), capsules, orally under moderate fat conditions on Day 1 in third intervention period; further followed by GSK3640254 200 mg (Treatment B- Test), tablets, orally under moderate fat conditions on Day 1 in first intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet; Drug: GSK3640254 Capsule
- Sequence 4 - Treatment DCBA (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment D- Test), tablets, orally under high fat conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment C- Reference), tablets, orally under fasted conditions on Day 1 in second intervention period; followed by GSK3640254 200 mg (Treatment B- Test), tablets, orally under moderate fat conditions on Day 1 in third intervention period; further followed by GSK3640254 200 mg (Treatment A- Reference), capsules, orally under moderate fat conditions on Day 1 in first intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet; Drug: GSK3640254 Capsule

INTERVENTIONS:
Drug: GSK3640254 Tablet — GSK3640254 tablets will contain mesylate salt with a unit dose of 100 mg (2x100 mg) and will be administered orally.
Drug: GSK3640254 Capsule — GSK3640254 capsules will contain mesylate salt with a unit dose of 100 mg (2x100 mg) and will be administered orally.

SUMMARY:
This is an open-label, single-dose, four-period, four sequential, and crossover study conducted to assess the relative bioavailability of GSK3640254 mesylate tablets and GSK3640254 mesylate capsules (in the presence of a moderate fat meal). This study will also evaluate the effect of food (fasted, moderate fat meal, and high fat meal) on the pharmacokinetics of GSK3640254 mesylate tablet formulation. Participants will be randomized to receive a single dose of GSK3640254 200 milligram (mg) capsules under moderate fat conditions and GSK3640254 200 mg tablets under moderate fat, fasted and high fat conditions in each treatment period. Approximately 16 participants will be enrolled and the duration of the study will be approximately 54 days.

ELIGIBILITY:
Inclusion Criteria

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Body weight >=50.0 kilogram (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 31.0 kg per square meter (m^2) (inclusive).
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male or female: Female participants: 1. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies: a. not a woman of childbearing potential (WOCBP); or Is a WOCBP and using a nonhormonal contraceptive method that is highly effective, with a failure rate of <1 percent (%), for 28 days before intervention, during the intervention period, and for at least 28 days after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. 2. A WOCBP must have a negative highly sensitive serum pregnancy test at Screening and Day -1. 3. Additional requirements for pregnancy testing during and after study intervention.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions.

Exclusion Criteria

* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal gastrointestinal (GI) anatomy or motility (example [e.g.], gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study intervention or render the participant unable to take oral study intervention.
* Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* Presence of hepatitis B surface antigen at Screening or within 3 months prior to starting study intervention.
* Positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention and positive on reflex to hepatitis C ribonucleic acid.
* Positive Human immunodeficiency virus-1 and -2 antigen/antibody immunoassay at Screening.
* ALT >1.5 × upper limit of normal (ULN). A single repeat of ALT is allowed within a single Screening period to determine eligibility.
* Bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
* Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of creatine phosphokinase and lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT, will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
* A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at Screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or non-prescription drugs including vitamins, herbal and dietary supplements (including Saint John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia Suicide Severity Rating Scale (C-SSRS).
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non sustained or sustained ventricular tachycardia, second degree atrioventricular block Mobitz Type II, third degree atrioventricular block, complete heart block, or conduction abnormality) which, in the opinion of the investigator or Medical Monitor, will interfere with the safety for the individual participant.
* Exclusion criteria for Screening ECG (a single repeat is allowed for eligibility determination): Heart rate: male <45 or >100 beats per minute (bpm) and female <50 or >100 bpm, and QTcF interval: male >450 millisecond (ms), female >450 ms.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 units. One unit is equivalent to 8 grams of alcohol: a half pint (~240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Unable to refrain from tobacco or nicotine-containing products within 3 months prior to Screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, open-label, single dose, 4 period crossover study in healthy participants conducted at a single center in the United States.
Pre-assignment Details: A total of 16 participants were enrolled in this study. The study was early terminated by sponsor due to a potential contamination issue in the study drug after completion of treatment Period 2. Hence, treatment Periods 3 and 4 were not conducted.
Groups:
- Sequence 1 - Treatment ABCD: Participants received a single dose of GSK3640254 200 mg capsules, orally under moderate fat conditions (Treatment A-reference) on Day 1 in treatment Period 1; followed by a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment B-test) on Day 1 in treatment Period 2. There was a washout period of at least 7 days between two treatment periods. Participants were planned to receive a single dose of GSK3640254 200 mg tablets, orally under fasted conditions (Treatment C-reference) on Day 1 in treatment Period 3; and a single dose of GSK3640254 200 mg tablets, orally under high fat conditions (Treatment D-test) on Day 1 in treatment Period 4. Treatment Periods 3 and 4 were planned but no participants were enrolled due to early termination of the study.
- Sequence 2 - Treatment BADC: Participants received a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment B-Test) on Day 1 in treatment Period 1; followed by a single dose of GSK3640254 200 mg capsules, orally under moderate fat conditions (Treatment A-Reference) on Day 1 in treatment Period 2. There was a washout period of at least 7 days between two treatment periods. Participants were planned to receive a single dose of GSK3640254 200 mg tablets, orally under high fat conditions (Treatment D-Test) on Day 1 in treatment Period 3; and a single dose of GSK3640254 200 mg tablets, orally under fasted conditions (Treatment C-Reference) on Day 1 in treatment Period 4. The treatment Periods 3 and 4 were planned but no participants were enrolled due to early termination of the study.
- Sequence 3 - Treatment CDAB: Participants received a single dose of GSK3640254 200 mg tablets, orally under fasted conditions (Treatment C-Reference) on Day 1 in treatment Period 1; followed by a single dose of GSK3640254 200 mg tablets, orally under high fat conditions (Treatment D-Test) on Day 1 in treatment Period 2. There was a washout period of at least 7 days between 2 treatment periods. Participants were planned to receive a single dose of GSK3640254 200 mg capsules, orally under moderate fat conditions (Treatment A-Reference) on Day 1 in treatment Period 3; and a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment B-Test) on Day 1 in treatment Period 4. The treatment Periods 3 and 4 were planned but no participants were enrolled due to early termination of the study.
- Sequence 4 - Treatment DCBA: Participants received a single dose of GSK3640254 200 mg tablets, orally under high fat conditions (Treatment D-Test) on Day 1 in treatment Period 1; followed by a single dose of GSK3640254 200 mg tablets, orally under fasted conditions (Treatment C-Reference) on Day 1 in treatment Period 2. There was a washout period of at least 7 days between 2 treatment periods. Participants were planned to receive a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment B-Test) on Day 1 in treatment Period 3; and a single dose of GSK3640254 200 mg capsules, orally under moderate fat conditions (Treatment A-Reference) on Day 1 in treatment Period 4. The treatment Periods 3 and 4 were planned but no participants were enrolled due to early termination of the study.
Period: Treatment Period 1 (1 Day)
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (Up to 7 Days)
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (1 Day)
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (Up to 7 Days)
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA
Started | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 4 | 4
Not completed — Study Closed/Terminated | 4 | 4 | 4 | 4
Period: Treatment Period 3 (1 Day)
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (Up to 7 Days)
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4 (1 Day)
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 - Treatment ABCD | Sequence 2 - Treatment BADC | Sequence 3 - Treatment CDAB | Sequence 4 - Treatment DCBA | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (8.46) | 33.8 (10.21) | 31.3 (7.68) | 38.0 (11.66) | 34.2 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2
  Male | 4 | 4 | 3 | 3 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 4 | 2 | 2 | 10
  White-White/Caucasian/European Heritage | 2 | 0 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC[0-infinity]) for GSK3640254 200 mg Capsules and Tablets Under Fed Condition (Treatment A and B)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis. PK Parameter Population included all participants who underwent plasma PK sampling and had evaluable PK parameters estimated.
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Treatment A- GSK3640254 200 mg Capsules (Fed): Participants received a single dose of GSK3640254 200 mg capsules, orally under moderate fat conditions (Treatment A-reference) on Day 1 in treatment Period 1 or 2.
- Treatment B- GSK3640254 200 mg Tablet (Fed): Participants received a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment B-test) on Day 1 in treatment Period 1 or 2.
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed)
Number analyzed (Participants) | 8 | 8
Hours*microgram per milliliter | 35.51 (16.7) | 31.16 (37.4)
Statistical Analysis 1: Comparison: Treatment A- GSK3640254 200 mg Capsules (Fed) vs Treatment B- GSK3640254 200 mg Tablet (Fed); Test type: Other; Ratio of Geometric Least Square Mean = 0.877, 90% CI 2-sided [0.7585 to 1.0152] — Relative bioavailability between treatment A and B assessed using analysis of variance with treatment, period, and sequence as fixed effects, participant as a random effect was performed on the natural log-transformed parameter of AUC(0-infinity)

2. Primary Outcome: AUC(0-infinity) for GSK3640254 200 mg Tablets Under Fasted and High Fat Condition (Treatment C and D)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Treatment C- GSK3640254 200 mg Tablet (Fasted): Participants received a single dose of GSK3640254 200 mg tablets, orally under fasted conditions (Treatment C-reference) on Day 1 in treatment Period 1 or 2.
- Treatment D- GSK3640254 200 mg Tablet (High Fat): Participants received a single dose of GSK3640254 200 mg tablets, orally under high fat conditions (Treatment D-test) on Day 1 in treatment Period 1 or 2.
Arm/Group | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 6 | 8
Hours*microgram per milliliter | 15.54 (49.4) | 37.85 (30.1)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time t (AUC[0-t]) for GSK3640254 200 mg Capsules and Tablets Under Fed Condition (Treatment A and B)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed)
Number analyzed (Participants) | 8 | 8
Hours*microgram per milliliter | 33.05 (18.2) | 29.50 (37.7)
Statistical Analysis 1: Comparison: Treatment A- GSK3640254 200 mg Capsules (Fed) vs Treatment B- GSK3640254 200 mg Tablet (Fed); Test type: Other; Ratio of Geometric Least Square Mean = 0.892, 90% CI 2-sided [0.7778 to 1.0239] — Relative bioavailability between treatment A and B assessed using analysis of variance with treatment, period, and sequence as fixed effects, participant as a random effect was performed on the natural log-transformed parameter of AUC(0-t)

4. Primary Outcome: AUC(0-t) for GSK3640254 200 mg Tablets Under Fasted and High Fat Condition (Treatment C and D)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 6 | 8
Hours*microgram per milliliter | 14.43 (52.3) | 34.99 (29.1)

5. Primary Outcome: Maximum Observed Concentration (Cmax) for GSK3640254 200 mg Capsules and Tablets Under Fed Condition (Treatment A and B)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed)
Number analyzed (Participants) | 8 | 8
Microgram per milliliter | 1.151 (16.8) | 1.088 (23.3)
Statistical Analysis 1: Comparison: Treatment A- GSK3640254 200 mg Capsules (Fed) vs Treatment B- GSK3640254 200 mg Tablet (Fed); Test type: Other; Ratio of Geometric Least Square Mean = 0.946, 90% CI 2-sided [0.8594 to 1.0404] — Relative bioavailability between treatment A and B assessed using analysis of variance with treatment, period, and sequence as fixed effects, participant as a random effect was performed on the natural log-transformed parameter of Cmax

6. Primary Outcome: Cmax for GSK3640254 200 mg Tablets Under Fasted and High Fat Condition (Treatment C and D)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 6 | 8
Microgram per milliliter | 0.5557 (71.3) | 1.168 (30.0)

7. Primary Outcome: Time of Cmax (Tmax) for GSK3640254 200 mg Capsules Under Fed Condition (Treatment A)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed)
Number analyzed (Participants) | 8
Hours | 6.000 [4.50 to 8.03]

8. Primary Outcome: Time of Cmax (Tmax) for GSK3640254 200 mg Tablets Under Fed, Fasted and High Fat Condition (Treatment B, C and D)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 6 | 8
Hours | 5.033 [3.00 to 6.07] | 4.250 [2.50 to 6.00] | 4.500 [2.00 to 12.00]
Statistical Analysis 1: Comparison: Treatment B- GSK3640254 200 mg Tablet (Fed) vs Treatment C- GSK3640254 200 mg Tablet (Fasted); Test type: Other; p = 0.4252, Wilcoxon signed-rank test — The p-value was assessed based on the Wilcoxon signed-rank test; Median Difference (Final Values) = 0.533, 90% CI 2-sided [-1.0000 to 2.0000] — The median difference and the 90 percent (%) confidence interval of the median difference was estimated from Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Treatment C- GSK3640254 200 mg Tablet (Fasted) vs Treatment D- GSK3640254 200 mg Tablet (High Fat); Test type: Other; p = 0.3125, Wilcoxon rank sum test — The p-value was assessed based on the Wilcoxon rank sum test; Median Difference (Final Values) = 1.000, 90% CI 2-sided [-0.7500 to 5.2500] — The median difference and the 90% confidence interval of the median difference were estimated from Hodges-Lehmann estimate

9. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; and other important medical events which may require medical or surgical intervention. Safety Population consisted of all participants who received at least 1 dose of study medication.
Time Frame: Up to Day 14
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  Any AEs | 0 | 1 | 0 | 1
  Any SAEs | 0 | 0 | 0 | 0

10. Secondary Outcome: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelet count.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
10^9 cells per liter
  Basophils | 0.024 (0.0092) | 0.028 (0.0175) | 0.036 (0.0119) | 0.038 (0.0139)
  Eosinophils | 0.086 (0.0472) | 0.096 (0.0910) | 0.126 (0.0761) | 0.128 (0.0740)
  Lymphocytes | 1.673 (0.3314) | 1.689 (0.2283) | 1.890 (0.4366) | 1.753 (0.4307)
  Monocytes | 0.365 (0.0849) | 0.384 (0.0968) | 0.434 (0.1492) | 0.410 (0.1610)
  Neutrophils | 2.324 (0.6459) | 2.403 (0.6452) | 2.470 (0.6709) | 2.403 (0.6713)
  Platelet count | 252.1 (22.64) | 241.5 (28.91) | 271.8 (44.08) | 270.9 (40.47)

11. Secondary Outcome: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Grams per liter | 145.1 (8.61) | 143.1 (8.63) | 144.8 (14.50) | 145.5 (12.81)

12. Secondary Outcome: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Proportion of red blood cells in blood | 0.4406 (0.02272) | 0.4344 (0.02477) | 0.4294 (0.04147) | 0.4345 (0.03691)

13. Secondary Outcome: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
10^12 cells per liter | 5.199 (0.3468) | 5.120 (0.3829) | 5.013 (0.5337) | 5.066 (0.4719)

14. Secondary Outcome: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Femtoliter | 84.88 (4.055) | 85.00 (4.184) | 85.84 (4.373) | 85.90 (4.178)

15. Secondary Outcome: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Picograms | 28.01 (1.864) | 28.06 (1.905) | 28.94 (1.614) | 28.73 (1.424)

16. Secondary Outcome: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and blood urea nitrogen.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Millimoles per liter
  Glucose | 4.774 (0.2447) | 4.780 (0.1336) | 4.843 (0.3617) | 4.838 (0.2467)
  Cholesterol | 4.853 (1.0266) | 4.630 (0.8081) | 5.028 (1.5207) | 4.960 (1.3009)
  Triglycerides | 1.048 (0.5887) | 0.989 (0.6469) | 1.509 (1.1537) | 1.379 (0.8660)
  Anion gap | 9.8 (1.58) | 9.9 (1.25) | 11.1 (2.03) | 10.9 (1.64)
  Calcium | 2.473 (0.0453) | 2.430 (0.0609) | 2.421 (0.1025) | 2.431 (0.1005)
  Carbon dioxide | 31.8 (1.16) | 31.3 (1.04) | 30.1 (2.30) | 30.5 (1.93)
  Chloride | 101.1 (0.99) | 101.0 (1.60) | 101.5 (2.14) | 101.6 (1.92)
  Phosphate | 1.173 (0.1278) | 1.201 (0.0606) | 1.199 (0.1929) | 1.230 (0.1292)
  Potassium | 4.56 (0.334) | 4.50 (0.239) | 4.28 (0.282) | 4.36 (0.272)
  Sodium | 138.1 (0.99) | 137.5 (2.00) | 138.5 (1.31) | 138.4 (1.19)
  Blood urea nitrogen | 4.785 (0.9271) | 4.509 (1.1031) | 4.351 (1.0179) | 4.096 (0.8941)

17. Secondary Outcome: Absolute Values for Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
International units per liter
  Creatine kinase | 116.1 (36.01) | 116.8 (48.18) | 94.8 (44.83) | 111.9 (55.35)
  Lactate dehydrogenase | 125.8 (9.54) | 122.1 (20.33) | 120.1 (18.18) | 122.3 (17.77)
  ALT | 18.1 (3.09) | 15.0 (3.46) | 17.9 (14.22) | 18.5 (15.32)
  ALP | 61.1 (8.89) | 58.3 (8.07) | 57.5 (14.82) | 60.8 (20.15)
  AST | 15.5 (2.39) | 14.4 (2.56) | 15.6 (3.11) | 16.1 (3.56)
  Gamma-glutamyl transferase | 18.3 (7.74) | 17.5 (7.54) | 28.4 (24.07) | 28.3 (21.26)

18. Secondary Outcome: Absolute Values for Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Micromoles per liter
  Urate | 289.9 (60.74) | 282.6 (60.69) | 287.0 (72.44) | 276.6 (60.99)
  Creatinine | 92.84 (12.612) | 92.71 (12.136) | 84.95 (13.200) | 82.78 (13.843)
  Bilirubin | 10.85 (2.838) | 10.78 (3.283) | 12.24 (5.172) | 11.09 (4.149)
  Direct bilirubin | 2.04 (0.526) | 2.13 (0.607) | 2.29 (1.241) | 2.14 (1.041)

19. Secondary Outcome: Absolute Values for Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Grams per liter
  Albumin | 45.8 (1.49) | 44.0 (1.77) | 45.9 (2.85) | 46.4 (3.20)
  Globulin | 27.8 (3.20) | 27.1 (4.02) | 25.3 (3.11) | 25.8 (2.92)
  Protein | 73.5 (2.56) | 71.1 (3.36) | 71.1 (3.98) | 72.1 (5.06)

20. Secondary Outcome: Absolute Values for Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Units per liter
  Amylase | 53.8 (11.51) | 54.3 (14.39) | 66.3 (26.29) | 68.8 (24.84)
  Lipase | 19.6 (10.00) | 21.6 (13.67) | 21.6 (11.69) | 22.9 (10.08)

21. Secondary Outcome: Absolute Values for Urine Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urine parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Ratio | 1.0169 (0.00666) | 1.0108 (0.00774) | 1.0165 (0.00590) | 1.0150 (0.00632)

22. Secondary Outcome: Absolute Values for Urine Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urine parameter: urobilinogen.
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Micromoles per liter | 3.3860 (0.00000) | 5.0790 (4.78853) | 8.4650 (7.00969) | 5.0790 (4.78853)

23. Secondary Outcome: Absolute Values for Urine Parameter: Potential of Hydrogen (pH)
Description: Urine samples were collected to analyze the urine parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0).
Time Frame: Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
pH | 6.38 (0.518) | 6.31 (0.704) | 6.31 (0.530) | 6.13 (0.641)

24. Secondary Outcome: Absolute Values for Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Fridericia's Formula (QTcF), Corrected QT Interval Using Bazett's Formula (QTcB)
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes.
Time Frame: Day 1: 2 hours and 4 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Milliseconds
  PR Interval: Day 1, 2 hours | 173.3 (9.62) | 173.4 (11.07) | 158.3 (17.85) | 156.9 (18.37)
  PR Interval: Day 1, 4 hours | 174.4 (11.25) | 173.0 (9.55) | 157.5 (14.29) | 149.6 (17.07)
  QRS Duration: Day 1, 2 hours | 90.9 (6.60) | 94.3 (6.02) | 91.5 (11.10) | 92.6 (10.68)
  QRS Duration: Day 1, 4 hours | 90.5 (5.88) | 91.4 (7.95) | 91.3 (9.13) | 92.1 (6.58)
  QT Interval: Day 1, 2 hours | 372.1 (22.03) | 372.8 (21.74) | 405.8 (25.73) | 387.6 (29.34)
  QT Interval: Day 1, 4 hours | 393.0 (22.55) | 391.0 (25.95) | 411.5 (30.29) | 398.3 (23.92)
  QTcF Interval: Day 1, 2 hours | 374.8 (14.41) | 376.0 (20.09) | 406.1 (23.12) | 399.9 (19.79)
  QTcF Interval: Day 1, 4 hours | 380.9 (18.00) | 381.1 (15.37) | 406.5 (24.60) | 410.6 (20.85)
  QTcB Interval: Day 1, 2 hours | 376.3 (13.54) | 377.9 (20.92) | 406.6 (26.45) | 406.8 (24.77)
  QTcB Interval: Day 1, 4 hours | 375.1 (18.55) | 376.5 (12.93) | 404.5 (28.43) | 417.4 (24.86)

25. Secondary Outcome: Absolute Values for Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without any distractions.
Time Frame: Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Millimeters of mercury
  SBP: Day 2 | 116.0 (8.05) | 115.1 (6.77) | 116.4 (10.25) | 118.3 (15.00)
  SBP: Day 3 | 116.4 (8.85) | 115.6 (10.34) | 117.1 (7.57) | 115.6 (9.66)
  SBP: Day 4 | 114.6 (8.45) | 117.6 (13.10) | 113.6 (11.33) | 116.5 (12.25)
  SBP: Day 5 | 113.4 (8.58) | 113.9 (10.58) | 113.8 (9.29) | 113.6 (7.01)
  DBP: Day 2 | 69.4 (6.61) | 69.6 (6.61) | 71.0 (8.16) | 71.0 (12.73)
  DBP: Day 3 | 65.3 (7.52) | 66.3 (9.75) | 68.6 (7.13) | 71.9 (9.28)
  DBP: Day 4 | 68.8 (9.71) | 68.9 (10.76) | 72.0 (9.38) | 73.4 (9.55)
  DBP: Day 5 | 70.0 (10.09) | 68.3 (11.65) | 72.4 (7.95) | 70.6 (6.70)

26. Secondary Outcome: Absolute Values for Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without any distractions.
Time Frame: Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Beats per minute
  Day 2 | 60.0 (6.19) | 61.3 (9.79) | 66.0 (11.75) | 64.5 (7.91)
  Day 3 | 62.5 (7.54) | 61.4 (9.07) | 63.4 (8.94) | 67.9 (9.57)
  Day 4 | 62.9 (9.51) | 61.9 (7.20) | 67.1 (8.39) | 64.5 (10.84)
  Day 5 | 60.4 (8.47) | 62.8 (11.21) | 67.4 (5.76) | 65.8 (9.27)

27. Secondary Outcome: Absolute Values for Respiratory Rate
Description: Respiratory rate was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Breaths per minute
  Day 2 | 14.3 (2.71) | 13.8 (2.25) | 14.0 (2.83) | 14.0 (3.55)
  Day 3 | 15.8 (1.98) | 15.5 (2.33) | 14.3 (1.98) | 14.3 (2.25)
  Day 4 | 16.0 (0.00) | 16.0 (1.07) | 14.5 (1.41) | 14.3 (2.25)
  Day 5 | 15.8 (3.62) | 15.3 (3.01) | 15.8 (2.25) | 14.5 (3.51)

28. Secondary Outcome: Absolute Values for Body Temperature
Description: Body temperature was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Degrees Celsius
  Day 2 | 36.15 (0.378) | 36.28 (0.292) | 36.15 (0.548) | 36.16 (0.407)
  Day 3 | 36.13 (0.219) | 36.34 (0.297) | 36.19 (0.230) | 36.11 (0.429)
  Day 4 | 36.21 (0.295) | 36.09 (0.242) | 36.26 (0.407) | 36.21 (0.253)
  Day 5 | 36.33 (0.238) | 36.41 (0.309) | 36.24 (0.213) | 36.36 (0.385)

29. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
10^9 cells per liter
  Basophils | -0.001 (0.0099) | 0.003 (0.0149) | -0.004 (0.0074) | -0.003 (0.0071)
  Eosinophils | -0.005 (0.0338) | 0.005 (0.0278) | 0.009 (0.0259) | 0.010 (0.0169)
  Lymphocytes | -0.170 (0.3945) | -0.154 (0.5025) | 0.015 (0.1927) | -0.123 (0.1959)
  Monocytes | -0.015 (0.0487) | 0.004 (0.0721) | 0.019 (0.0884) | -0.005 (0.0767)
  Neutrophils | -0.214 (0.4939) | -0.135 (0.2945) | -0.166 (0.7631) | -0.234 (0.5199)
  Platelet count | 18.3 (22.63) | 7.6 (11.84) | 6.1 (18.76) | 5.3 (18.38)

30. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Grams per liter | 6.0 (4.34) | 4.0 (4.93) | 3.3 (6.50) | 4.0 (7.33)

31. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Proportion of red blood cells in blood | 0.0179 (0.01374) | 0.0116 (0.01430) | 0.0063 (0.01884) | 0.0114 (0.01963)

32. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
10^12 cells per liter | 0.241 (0.1604) | 0.163 (0.1521) | 0.100 (0.2321) | 0.154 (0.2329)

33. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Femtoliter | -0.61 (0.416) | -0.49 (0.582) | -0.45 (0.672) | -0.39 (0.340)

34. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Picograms | -0.10 (0.245) | -0.05 (0.220) | 0.09 (0.387) | -0.13 (0.306)

35. Secondary Outcome: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and blood urea nitrogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Millimoles per liter
  Glucose | -0.055 (0.3778) | -0.049 (0.2568) | -0.168 (0.2530) | -0.173 (0.3159)
  Cholesterol | 0.498 (0.7449) | 0.275 (0.4277) | 0.310 (0.4079) | 0.243 (0.3383)
  Triglycerides | 0.026 (0.1434) | -0.033 (0.1849) | 0.013 (0.5576) | -0.118 (0.4461)
  Anion gap | -0.9 (1.89) | -0.8 (2.25) | -0.6 (1.41) | -0.9 (2.17)
  Calcium | 0.095 (0.0674) | 0.053 (0.0794) | 0.026 (0.0713) | 0.036 (0.0965)
  Carbon dioxide | 1.4 (1.19) | 0.9 (1.46) | 1.3 (0.89) | 1.6 (1.51)
  Chloride | 0.3 (1.49) | 0.1 (2.17) | -0.1 (1.25) | 0.0 (1.85)
  Phosphate | -0.006 (0.1165) | 0.023 (0.1499) | 0.044 (0.1327) | 0.075 (0.1144)
  Potassium | 0.33 (0.238) | 0.26 (0.226) | 0.08 (0.198) | 0.16 (0.239)
  Sodium | 0.4 (1.60) | -0.3 (2.25) | 0.4 (1.30) | 0.3 (1.58)
  Blood urea nitrogen | -0.049 (0.8640) | -0.325 (0.7951) | 0.090 (1.7057) | -0.165 (1.4390)

36. Secondary Outcome: Change From Baseline in Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
International units per liter
  Creatine kinase | -54.3 (60.14) | -53.6 (72.20) | -24.5 (24.18) | -7.4 (34.16)
  Lactate dehydrogenase | -9.6 (16.62) | -13.3 (19.02) | -12.9 (8.22) | -10.8 (7.81)
  ALT | 1.0 (2.56) | -2.1 (3.00) | 0.4 (2.50) | 1.0 (2.00)
  ALP | -0.9 (8.11) | -3.8 (4.77) | -3.0 (5.58) | 0.3 (3.73)
  AST | -1.1 (2.03) | -2.3 (2.38) | -0.5 (1.07) | 0.0 (2.73)
  Gamma-glutamyl transferase | 1.4 (2.13) | 0.6 (1.77) | -1.1 (1.46) | -1.3 (6.45)

37. Secondary Outcome: Change From Baseline in Chemistry Parameters: Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Micromoles per liter
  Urate | -6.3 (18.71) | -13.5 (28.10) | -14.1 (37.84) | -24.5 (50.08)
  Creatinine | 1.66 (6.736) | 1.54 (6.292) | 1.75 (8.188) | -0.43 (7.123)
  Bilirubin | 3.13 (2.364) | 3.05 (2.117) | 1.13 (4.318) | -0.03 (4.639)
  Direct bilirubin | 0.43 (0.590) | 0.51 (0.449) | 0.06 (0.609) | -0.09 (0.762)

38. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Grams per liter
  Albumin | 1.5 (2.83) | -0.3 (2.38) | 0.1 (1.55) | 0.6 (2.67)
  Globulin | 0.5 (1.85) | -0.1 (2.30) | -0.4 (2.13) | 0.1 (2.42)
  Protein | 2.0 (4.60) | -0.4 (3.78) | -0.3 (2.87) | 0.8 (4.77)

39. Secondary Outcome: Change From Baseline in Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Units per liter
  Amylase | 1.0 (9.29) | 1.5 (10.21) | 4.0 (5.98) | 6.5 (6.32)
  Lipase | -9.5 (16.34) | -7.5 (9.93) | -3.9 (3.87) | -2.6 (6.25)

40. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Ratio | 0.0034 (0.01006) | -0.0028 (0.01341) | -0.0009 (0.01284) | -0.0024 (0.01097)

41. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Micromoles per liter | -1.6930 (4.78853) | 0.0000 (7.23957) | 1.6930 (8.67994) | -1.6930 (4.78853)

42. Secondary Outcome: Change From Baseline in Urinalysis Parameter: pH
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, prior to the first dose of study drug administration. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
pH | 0.25 (0.463) | 0.19 (0.651) | 0.44 (0.623) | 0.25 (0.926)

43. Secondary Outcome: Change From Baseline in PR Interval, QRS Duration, QT Interval, QTcF, QTcB
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes. Baseline was defined as the average of the triplicate pre-dose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 hours and 4 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Milliseconds
  PR Interval: Day 1, 2 hours | -6.3 (3.81) | 2.3 (8.24) | -0.3 (5.85) | 5.4 (14.35)
  PR Interval: Day 1, 4 hours | -5.1 (4.79) | 1.9 (6.24) | -1.0 (7.21) | -1.9 (15.87)
  QRS Duration: Day 1, 2 hours | 1.4 (3.81) | 3.5 (6.74) | 0.3 (4.46) | 1.6 (5.29)
  QRS Duration: Day 1, 4 hours | 1.0 (5.37) | 0.6 (4.44) | 0.0 (4.44) | 1.1 (3.14)
  QT Interval: Day 1, 2 hours | -10.9 (11.37) | -15.6 (12.64) | 5.5 (7.96) | -12.6 (13.98)
  QT Interval: Day 1, 4 hours | 10.0 (16.40) | 2.6 (10.69) | 11.3 (13.72) | -2.0 (15.30)
  QTcF Interval: Day 1, 2 hours | -6.9 (8.92) | -10.5 (6.57) | -0.1 (6.36) | -7.5 (8.00)
  QTcF Interval: Day 1, 4 hours | -0.8 (11.34) | -5.4 (6.67) | 0.3 (7.74) | 3.3 (4.89)
  QTcB Interval: Day 1, 2 hours | -4.8 (14.38) | -8.1 (13.15) | -3.1 (8.79) | -4.6 (11.84)
  QTcB Interval: Day 1, 4 hours | -5.9 (16.44) | -9.5 (9.81) | -5.3 (11.66) | 6.0 (5.37)

44. Secondary Outcome: Change From Baseline in SBP and DBP
Description: SBP and DBP were measured in the semi-recumbent position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without any distractions. Baseline was defined as the average of the triplicate pre-dose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Millimeters of mercury
  SBP: Day 2 | -0.1 (3.87) | -2.0 (4.54) | -1.8 (6.94) | 3.4 (10.42)
  SBP: Day 3 | 0.3 (3.20) | -1.5 (7.31) | -1.0 (6.70) | 0.8 (4.74)
  SBP: Day 4 | -1.5 (8.96) | 0.5 (9.21) | -4.5 (7.54) | 1.6 (6.59)
  SBP: Day 5 | -2.8 (6.41) | -3.3 (7.09) | -4.4 (9.29) | -1.3 (6.36)
  DBP: Day 2 | -2.3 (4.65) | -3.0 (6.50) | -1.9 (4.55) | -0.9 (6.56)
  DBP: Day 3 | -6.4 (7.98) | -6.4 (5.78) | -4.3 (4.83) | 0.0 (3.38)
  DBP: Day 4 | -2.9 (7.00) | -3.8 (7.76) | -0.9 (6.53) | 1.5 (5.78)
  DBP: Day 5 | -1.6 (4.75) | -4.4 (7.56) | -0.5 (4.69) | -1.3 (5.28)

45. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the semi-recumbent position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without any distractions. Baseline was defined as the average of the triplicate pre-dose assessments within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Beats per minute
  Day 2 | -2.0 (4.84) | -0.6 (6.67) | 1.4 (6.95) | 1.4 (3.85)
  Day 3 | 0.5 (6.07) | -0.5 (4.38) | -1.3 (5.55) | 4.8 (5.97)
  Day 4 | 0.9 (5.44) | 0.0 (7.93) | 2.5 (4.34) | 1.4 (6.25)
  Day 5 | -1.6 (5.60) | 0.9 (4.94) | 2.8 (3.20) | 2.6 (7.85)

46. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Breaths per minute
  Day 2 | -0.3 (4.83) | 0.3 (2.71) | -0.5 (2.33) | 0.3 (3.62)
  Day 3 | 1.3 (2.12) | 2.0 (3.21) | -0.3 (1.98) | 0.5 (2.56)
  Day 4 | 1.5 (2.56) | 2.5 (2.07) | 0.0 (2.14) | 0.5 (3.16)
  Day 5 | 1.3 (5.65) | 1.8 (4.06) | 1.3 (1.83) | 0.8 (3.37)

47. Secondary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured in the semi-recumbent position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose), Days 2, 3, 4, and 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Degrees Celsius
  Day 2 | -0.10 (0.374) | -0.10 (0.227) | -0.15 (0.469) | -0.10 (0.417)
  Day 3 | -0.13 (0.433) | -0.04 (0.311) | -0.11 (0.253) | -0.15 (0.389)
  Day 4 | -0.04 (0.262) | -0.29 (0.429) | -0.04 (0.450) | -0.05 (0.288)
  Day 5 | 0.08 (0.354) | 0.04 (0.256) | -0.06 (0.250) | 0.10 (0.342)

48. Secondary Outcome: Lag Time for Absorption (Tlag) for GSK3640254
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 6 | 8
Hours | 0.000 [0.00 to 2.00] | 0.000 [0.00 to 1.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]

49. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) for GSK3640254
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 6 | 8
Hours | 23.607 (18.7) | 22.001 (12.3) | 22.948 (29.2) | 24.448 (22.3)

50. Secondary Outcome: Apparent Oral Clearance (CL/F) for GSK3640254
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 6 | 8
Liters per hour | 5.632 (16.7) | 6.418 (37.4) | 12.87 (49.4) | 5.284 (30.1)

51. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for GSK3640254
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 6 | 8
Liters | 191.8 (30.8) | 203.7 (42.7) | 426.1 (70.7) | 186.4 (33.5)

52. Secondary Outcome: Plasma Pharmacokinetic Concentration of GSK3640254
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The PK Concentration Population included all participants who underwent plasma PK sampling and had evaluable PK assay results.
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Concentration Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 8 | 8 | 6 | 8
Nanogram per milliliter
  Pre-dose | NA (NA) — Mean could not be calculated as it was below the limit of quantification; standard deviation (SD) could not be calculated due to the high proportion of NQ values (>30% of values were imputed i.e. NQ assigned zero concentration) which affected the SD. | 7.863 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 3.227 (NA) — Standard deviation could not be calculated due to high proportion of NQ values (>30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | NA (NA) — Mean could not be calculated as it was below the limit of quantification; standard deviation (SD) could not be calculated due to the high proportion of NQ values (>30% of values were imputed i.e. NQ assigned zero concentration) which affected the SD.
  1 hour | 14.83 (NA) — Standard deviation could not be calculated due to high proportion of NQ values (>30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation | 68.15 (70.107) | 61.22 (75.133) | 443.0 (456.37)
  1.5 hours | 62.30 (87.234) | 291.1 (304.32) | 145.5 (121.20) | 696.0 (627.36)
  2 hours | 148.5 (176.30) | 486.0 (352.74) | 273.2 (206.53) | 837.6 (602.91)
  2.5 hours | 293.4 (267.01) | 746.1 (448.03) | 371.0 (261.44) | 946.3 (477.31)
  3 hours | 490.3 (384.97) | 893.4 (398.47) | 412.4 (286.00) | 1009 (402.66)
  3.5 hours | 647.1 (375.90) | 926.3 (194.74) | 477.2 (345.06) | 976.3 (339.08)
  4 hours | 759.3 (334.79) | 955.8 (253.23) | 541.0 (463.54) | 1024 (350.97)
  4.5 hours | 919.1 (287.70) | 1027 (320.44) | 624.0 (475.10) | 1027 (290.12)
  5 hours | 1057 (172.77) | 1024 (278.55) | 560.3 (407.61) | 1067 (321.21)
  6 hours | 1129 (204.39) | 1006 (231.01) | 523.5 (319.40) | 1001 (245.94)
  8 hours | 1020 (201.61) | 890.6 (277.11) | 471.8 (294.06) | 922.1 (238.72)
  12 hours | 793.1 (134.74) | 713.6 (247.97) | 359.5 (226.80) | 795.3 (206.96)
  24 hours | 581.8 (156.89) | 519.8 (184.90) | 262.7 (140.32) | 597.5 (175.90)
  48 hours | 268.0 (52.285) | 240.5 (84.134) | 124.2 (50.302) | 281.6 (75.989)
  72 hours | 131.0 (26.340) | 116.5 (38.362) | 56.97 (16.732) | 147.8 (56.122)
  96 hours | 67.26 (18.506) | 52.96 (17.846) | 28.18 (11.700) | 78.38 (39.314)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from start of the treatment (Day 1) up to Day 14
Description: Safety Population consisted of all participants who received at least 1 dose of study medication. Data is presented for Periods 1 and 2 only as data was not collected in Periods 3 and 4 due to early termination of the study following completion of Period 2.
Arm/Group | Treatment A- GSK3640254 200 mg Capsules (Fed) | Treatment B- GSK3640254 200 mg Tablet (Fed) | Treatment C- GSK3640254 200 mg Tablet (Fasted) | Treatment D- GSK3640254 200 mg Tablet (High Fat)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A- GSK3640254 200 mg Capsules (Fed) (N=8) | Treatment B- GSK3640254 200 mg Tablet (Fed) (N=8) | Treatment C- GSK3640254 200 mg Tablet (Fasted) (N=8) | Treatment D- GSK3640254 200 mg Tablet (High Fat) (N=8)
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT04128293/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04128293/SAP_001.pdf